CLINICAL TRIAL: NCT03065712
Title: Test - Retest Reproducibility of 18F Fluoroestradiol (FES) PET and Predictive Measure for Endocrine Therapy Response in Patients With Newly Diagnosed Metastatic Breast Cancer
Brief Title: Test - Retest Reproducibility of 18F Fluoroestradiol (FES) PET
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Competing clinical trial
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STU 032016-021
Record Dates: First submitted 2017-02-20; First posted 2017-02-28 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2019-08

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; PET/CT; FES; 18F Fluoroestradiol; Breast
MeSH Terms: conditions — Breast Neoplasms | interventions — 16-fluoroestradiol; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FES PET/CT (Experimental): This is a single arm study that involves FES PET/CT.
  Procedure: Computed Tomography
  * Drug: [F-18] fluoroestradiol: [F-18]FES
  * Other: Laboratory Biomarker Analysis
  * Procedure: Positron Emission Tomography
  Interventions: Drug: F-18 Fluoroestradiol; Procedure: Computed Tomography; Procedure: Positron Emission Tomography; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: F-18 Fluoroestradiol — F-18 Fluoroestradiol will be administered for PET/CT scan.
  Other Names: FES PET/CT; F-18 Fluoroestradiol PET/CT
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; CT Scan
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; positron emission tomography scan; Positron-Emission Tomography
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This study will formally address the hypothesis that FES-PET/CT measurement of ER expression predicts clinical benefit of first-line endocrine therapy in newly diagnosed ER+ metastatic breast cancer patients and establishes the repeatability of FES PET/CT.

DETAILED DESCRIPTION:
The experimental FES-PET/CT is required to be completed 0 to 30 days prior to initiation of first-line endocrine therapy for metastatic ER+ breast cancer. Labs and correlative radiology, as directed per clinical care, are required within 60 days prior to FES-PET/CT; and FDG-PET/CT is required within 60 days before the FES-PET/CT. Follow-up will comprise 24 months of standard practice treatment and follow up.

Visit 1: Patients will have at least one visit with investigator (or investigator designee) prior to the study to review clinical history and prior treatment of primary breast cancer, and to explain the study. Correlative radiology studies including CT, MRI, or bone scan as per institutional routine clinical care, and any clinically-directed laboratory tests performed as part of metastatic staging must be performed within 60 days of the FES-PET/CT.

Visit 2: The patient will have a clinically-directed FDG-PET/CT as part of metastatic staging. The FDG-PET/CT will usually be obtained within 60 days prior to the FES-PET/CT. It may be done up to 30 days before the FES-PET/CT if there has been no endocrine therapy for metastatic disease started before the FES-PET/CT. The FDG-PET/CT and FES-PET/CT cannot be performed on the same day due to the half-life of F-18. The FDG-PET/CT may be done as a research scan, if the patient is unable to obtain a clinically-directed FDG-PET/CT as part of their clinical care or within 60 days of FES PET/CT. The research FDG-PET/CT, in this instance, will be identical in procedure to the institution's clinical FDG-PET/CT. The blood glucose level will be < 200 mg/dl, before FDG injection, which is institutional standard clinical protocol. The following additional patient data will be obtained: histological diagnosis of primary and/or metastatic disease, date of diagnosis of primary and metastatic disease, gender, height, weight (for BMI), ECOG score, and prior adjuvant and metastatic treatment regimens used.

Visit 3 - Day of FES PET/CT: The patient will have an intravenous line placed typically in the hand or arm opposite to the known primary breast cancer, FES will be given by 2 minute infusion, and the dose administered will be approximately 6mCi +/- 20%. After approximately 60+/- 10 minutes of uptake time, the patient will be positioned supine in the PET/CT scanner for standard whole body PET/CT scan from the skull base to mid-thigh. This scan will take approximately 20-30 min. If there are any breast lesions, a higher resolution PEM study of the breast/s may be obtained which make take approximately an additional 30-60 min.

A blood sample to be obtained, just before the FES injection, and submitted for hormonal analysis (estradiol and sex hormone binding globulin).

Visit 4-Day of Reproducibility FES-PET/CT: The test re-test FES-PET/CT will need to be performed at least 24 hours after the first FES-PET/CT and no later than 10 days following the initial FES study, and it can be done at any time after the FDG-PET/CT. The second FES-PET/CT study must be performed on the same scanner as the first FES-PET/CT and the imaging protocol described in Visit 3 should be closely followed. If there are any breast lesions, a higher resolution PEM study may be obtained which make take approximately an additional 30 min.

Visit 5-Week 1 to 4 after first FES-PET/CT: Patients will start endocrine therapy in the period from 0 to 30 days post FES-PET/CT, as per clinical standard.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be over 18 years old and capable and willing to provide informed consent.
* Patients of childbearing potential must have a negative urine or serum pregnancy test within 7 days prior to PET/CT imaging per institution's standard of care;
* A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria;
* Has not undergone a hysterectomy or bilateral oophorectomy; or
* Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
* Medically stable as judged by patient's physician.
* Life expectancy must be estimated at > 6 months.
* Patients must have an ECOG performance status of 0-3 (restricted to ECOG PS 0-2 if age >70 years).
* Patients with known allergic or hypersensitivity reactions to previously administered radiopharmaceuticals of similar chemical or biologic composition to FES are NOT eligible.
* Patients with liver failure are NOT eligible.
* Patient must NOT be breast-feeding.
* Histologically confirmed ER+ breast cancer either from a metastatic biopsy or from a primary breast tumor with imaging evidence of metastatic disease. The pathology report and either (1) tumor tissue (blocks or unstained slides) or (2) a photomicrograph of the ER IHC slide from at least one site of metastatic disease
* No prior endocrine therapy for metastatic disease is allowed (i.e. must be first-line endocrine therapy for metastatic disease). However, a history of adjuvant endocrine therapy is allowed, as long as the date of diagnosis of metastatic disease is > 2 years following initiation of adjuvant endocrine therapy. Patients who develop metastatic disease while still receiving adjuvant endocrine therapy must have a change in the type of endocrine agent used for subsequent metastatic disease treatment. Patients on blocking adjuvant therapy (with a blocking agent such as toremifene or tamoxifen) must be off the agents for a minimum of 60 days to allow for adequate uptake of FES
* Patients with human epidermal growth factor-2 positive (HER2+) metastatic tumors are NOT eligible
* Postmenopausal women, men, or premenopausal women for whom endocrine therapy (tamoxifen, aromatase inhibitor (AI) with or without ovarian suppression or fulvestrant), with or without a CDK4/6 inhibitor is planned after FES-PET/CT is completed
* Disease may be measurable (by RECIST 1.1 criteria) or non-measurable but must be present in at least one non-liver site, 1.5 cm or greater and visualized on PET/CT with [18F]-fluorodeoxyglucose (FDG). Patients with effusion only disease or disease only in the liver are not eligible for the study
* Patient must be able to lie still for a 20 to 30 minute PET/CT scan.

Exclusion Criteria:

. Patients not meeting the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2020-02-22 (Estimated); Study Completion 2021-02-20 (Estimated)

PRIMARY OUTCOMES:
Repeatablility coefficient | Repeatable FES PET/CT scans are performed within 10 days
  Maximum standardized uptake value repeatability coefficient

SECONDARY OUTCOMES:
Negative Predictive Value | 6 months after treatment completion
  Negative Predictive Value of baseline FES PET/CT

CONTACTS AND LOCATIONS:
Overall Officials: Rathan Subramaniam, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Clements University Hospital, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mintun MA, Welch MJ, Siegel BA, Mathias CJ, Brodack JW, McGuire AH, Katzenellenbogen JA. Breast cancer: PET imaging of estrogen receptors. Radiology. 1988 Oct;169(1):45-8. doi: 10.1148/radiology.169.1.3262228.
- [Background] Mortimer JE, Dehdashti F, Siegel BA, Trinkaus K, Katzenellenbogen JA, Welch MJ. Metabolic flare: indicator of hormone responsiveness in advanced breast cancer. J Clin Oncol. 2001 Jun 1;19(11):2797-803. doi: 10.1200/JCO.2001.19.11.2797. PMID 11387350
- [Background] Mortimer JE, Dehdashti F, Siegel BA, Katzenellenbogen JA, Fracasso P, Welch MJ. Positron emission tomography with 2-[18F]Fluoro-2-deoxy-D-glucose and 16alpha-[18F]fluoro-17beta-estradiol in breast cancer: correlation with estrogen receptor status and response to systemic therapy. Clin Cancer Res. 1996 Jun;2(6):933-9. PMID 9816253
- [Background] Linden HM, Stekhova SA, Link JM, Gralow JR, Livingston RB, Ellis GK, Petra PH, Peterson LM, Schubert EK, Dunnwald LK, Krohn KA, Mankoff DA. Quantitative fluoroestradiol positron emission tomography imaging predicts response to endocrine treatment in breast cancer. J Clin Oncol. 2006 Jun 20;24(18):2793-9. doi: 10.1200/JCO.2005.04.3810. Epub 2006 May 8. PMID 16682724
- [Background] Kurland BF, Peterson LM, Lee JH, Linden HM, Schubert EK, Dunnwald LK, Link JM, Krohn KA, Mankoff DA. Between-patient and within-patient (site-to-site) variability in estrogen receptor binding, measured in vivo by 18F-fluoroestradiol PET. J Nucl Med. 2011 Oct;52(10):1541-9. doi: 10.2967/jnumed.111.091439. Epub 2011 Sep 8. PMID 21903739
- [Background] Dehdashti F, Mortimer JE, Trinkaus K, Naughton MJ, Ellis M, Katzenellenbogen JA, Welch MJ, Siegel BA. PET-based estradiol challenge as a predictive biomarker of response to endocrine therapy in women with estrogen-receptor-positive breast cancer. Breast Cancer Res Treat. 2009 Feb;113(3):509-17. doi: 10.1007/s10549-008-9953-0. Epub 2008 Mar 9. PMID 18327670
- [Background] Linden HM, Kurland BF, Peterson LM, Schubert EK, Gralow JR, Specht JM, Ellis GK, Lawton TJ, Livingston RB, Petra PH, Link JM, Krohn KA, Mankoff DA. Fluoroestradiol positron emission tomography reveals differences in pharmacodynamics of aromatase inhibitors, tamoxifen, and fulvestrant in patients with metastatic breast cancer. Clin Cancer Res. 2011 Jul 15;17(14):4799-805. doi: 10.1158/1078-0432.CCR-10-3321. Epub 2011 Jul 12. PMID 21750198
- [Background] Peterson LM, Kurland BF, Schubert EK, Link JM, Gadi VK, Specht JM, Eary JF, Porter P, Shankar LK, Mankoff DA, Linden HM. A phase 2 study of 16alpha-[18F]-fluoro-17beta-estradiol positron emission tomography (FES-PET) as a marker of hormone sensitivity in metastatic breast cancer (MBC). Mol Imaging Biol. 2014 Jun;16(3):431-40. doi: 10.1007/s11307-013-0699-7. Epub 2013 Oct 30. PMID 24170452